CLINICAL TRIAL: NCT06850220
Title: Observational Study on the Impact of Obstructive Sleep Apnea on Executive Function and Empathy Development in Children
Acronym: OSA-EFED
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Ying Wu, Chief Physician, Children's Hospital of Soochow University
Other Study IDs: 2024005
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Obstructive Sleep Apnea; Cognition; Empathy; EEG
Keywords: Obstructive Sleep Apnea; Executive Function; Empathy; Children; EEG Biomarkers; Cohort Study; Neurodevelopment; Adenotonsillectomy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Mild OSA - Surgical Treatment Group: Children aged 3-12 years diagnosed with mild OSA (1 < OAHI ≤ 5 events/hour) who undergo adenotonsillectomy as the primary treatment.
- Mild OSA - Pharmacological Group: Children aged 3-12 years diagnosed with mild OSA (1 < OAHI ≤ 5 events/hour) who receive conservative treatment with nasal corticosteroids and leukotriene receptor antagonists.
- Moderate OSA Group: Children aged 3-12 years diagnosed with moderate OSA (5 < OAHI ≤ 10 events/hour) who undergo adenotonsillectomy as the primary treatment.
- Severe OSA Group: Children aged 3-12 years diagnosed with severe OSA (OAHI > 10 events/hour) who undergo adenotonsillectomy as the primary treatment.
- Healthy Control Group: Healthy children aged 3-12 years with no history of OSA or other sleep disorders. This group serves as a control for comparison.

SUMMARY:
This study aims to investigate the effects of obstructive sleep apnea (OSA) on executive function and empathy development in children aged 3-12 years. The study will compare the outcomes of different treatment approaches (surgical vs. pharmacological) in children with mild OSA and track the progression of cognitive and emotional functions over 12 months. The study will also explore potential EEG biomarkers for assessing neurological damage in OSA children.

DETAILED DESCRIPTION:
This is a prospective observational cohort study conducted at the Sleep Center of the Respiratory Department and the Department of Child and Adolescent Healthcare, Children's Hospital of Soochow University. Children diagnosed with OSA will be divided into groups based on disease severity (mild, moderate, severe) and treatment choice (surgical or pharmacological). The study will assess executive function and empathy levels at baseline, 6 months, and 12 months post-intervention using behavioral tests, EEG, and parent-reported questionnaires. The study aims to provide evidence for treatment selection in mild OSA children and identify EEG biomarkers for neurological damage.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-12 years.
* Diagnosed with OSA due to adenoid and/or tonsillar hypertrophy.
* IQ ≥ 85.
* Parental consent for participation.

Exclusion Criteria:

* Other primary sleep disorders (e.g., narcolepsy, restless leg syndrome).
* Developmental delay, epilepsy, or other neurological/metabolic disorders.
* Chronic diseases or history of head trauma.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 3-12 years diagnosed with OSA and healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Executive function measured by the "Heart and Flower" task. | Baseline, 6 months, and 12 months
  Children's executive function will be assessed using the "Heart and Flower" task, which measures the ability to follow rules and switch between tasks. Performance is evaluated based on accuracy and reaction time.
Empathy Level Measured by the Pain Empathy Paradigm | Baseline, 6 months, and 12 months
  Children's empathy level will be assessed using a pain empathy paradigm, where children rate the pain intensity of others in pictures. Scores reflect their ability to understand and share the feelings of others.
Parent-Reported Executive Function Using BRIEF-P Questionnaire | Baseline, 6 months, and 12 months
  Parents will complete the BRIEF-P to assess their child's everyday executive function behaviors, including inhibition, emotional control, and working memory.
Working Memory Assessed by WPPSI-IV or WISC-IV | Baseline, 6 months, and 12 months
  Children's working memory will be assessed using the WPPSI-IV or WISC-IV, depending on the child's age.

SECONDARY OUTCOMES:
Obstructive Apnea-Hypopnea Index (OAHI) Measured by PSG | Baseline, 6 months, and 12 months
  The OAHI, which measures the number of obstructive apnea and hypopnea events per hour during sleep, will be assessed using polysomnography (PSG).
Minimum Oxygen Saturation (MinSaO2) During Sleep | Baseline, 6 months, and 12 months
  The minimum oxygen saturation level during sleep will be measured using PSG to assess the severity of oxygen desaturation in OSA children.
Parent-Reported Sleep Habits Using CSHQ Questionnaire | Baseline, 6 months, and 12 months
  Parents will complete the CSHQ to report their child's sleep behaviors, including bedtime resistance, sleep duration, and night awakenings.
Theta Wave Intensity in Prefrontal Cortex During Executive Function Tasks | Baseline, 6 months, and 12 months
  EEG will be used to measure theta wave intensity in the prefrontal cortex while children perform executive function tasks, providing an objective neural correlate of executive function.

OTHER OUTCOMES:
Theta/Beta Ratio in Resting-State EEG | Baseline, 6 months, and 12 months
  The theta/beta ratio in resting-state EEG will be measured as a potential biomarker for cognitive and emotional regulation in children with OSA.
Event-Related Potentials (N2 and LPP) During Empathy Tasks | Baseline, 6 months, and 12 months
  EEG will be used to measure event-related potentials (N2 and LPP) during empathy tasks, reflecting neural responses to emotional stimuli.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant privacy and confidentiality, as the data contains sensitive information related to children's health and neuropsychological development.